CLINICAL TRIAL: NCT02125578
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled, Multiple-Dose, Dose-Ranging, Parallel-Group Study of PEGylated Interferon Beta-1a (BIIB017) in Healthy Volunteers
Brief Title: A Multiple Dose Safety Study of PEG-IFN in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 105HV102
Record Dates: First submitted 2014-04-25; First posted 2014-04-29 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- BIIB017 (PEGylated Interferon Beta-1a) (Experimental): Varying doses (63 mcg up to 188 mcg) of BIIB017 will be administered SC every other week for a total of 6 weeks.
  Interventions: Drug: BIIB017 (PEGylated Interferon Beta-1a)
- BIIB017 (PEGylated Interferon Beta-1a) and Placebo (Experimental): Varying doses (63 mcg up to 188 mcg) of BIIB017 will be administered SC every 4 weeks for a total of 6 weeks. To ensure blinding, each subject will receive placebo every other week.
  Interventions: Drug: BIIB017 (PEGylated Interferon Beta-1a); Drug: Placebo
- Placebo (Placebo Comparator): Placebo dose will be administered SC every other week for a total of 6 weeks.
  Interventions: Drug: BIIB017 (PEGylated Interferon Beta-1a)

INTERVENTIONS:
Drug: BIIB017 (PEGylated Interferon Beta-1a) — Each participant will receive BIIB017 every other week or every 4 weeks.
Drug: Placebo — Each participant will receive placebo every other week or every 4 weeks.
  Arms: BIIB017 (PEGylated Interferon Beta-1a) and Placebo

SUMMARY:
The primary objectives are to identify the highest safe and well-tolerated dose and frequency of BIIB017 (PEGylated Interferon Beta-1a) subcutaneous (SC), within the range of 63 to 188 mcg, when given every other week or every 4 weeks to healthy volunteers (HV).

ELIGIBILITY:
Key Inclusion Criteria:

* Body Mass Index (BMI) of 18 to 35 kg/m2, inclusive, and a minimum body weight of 50.0 kg at screening.
* All male subjects and female subjects of child-bearing potential must be willing and able to practice effective birth control during the study and be willing and able to continue contraception for 30 days after their last dose of study treatment.

Key Exclusion Criteria:

* Abnormal screening and baseline blood and urine tests determined to be clinically significant by the Investigator.
* Hematologic or hepatic enzyme laboratory values that were outside the normal range.
* History of severe allergic or anaphylactic reactions.
* History of any clinically-significant (as determined by the Investigator) cardiac, endocrinologic, hematologic, hepatic, immunologic, metabolic, urologic, pulmonary, neurologic, dermatologic, psychiatric, renal and/or other major disease, and/or history of seizure disorder.
* A family history of MS in a first-degree relative.
* A fever (body temperature >38°C) or symptomatic viral or bacterial infection (including upper respiratory infection) within 1 week prior to Day 1.
* Abnormal ECG values as determined by the Investigator.
* Positive test result for hepatitis C antibody, hepatitis B surface antigen (HBsAg), or human immunodeficiency virus (HIV) antibody.
* Female subjects who are considering pregnancy, currently pregnant or breastfeeding.
* Subjects who received a tattoo or body piercing (including earring) within 60 days of baseline or subjects who are considering getting a tattoo or body piercing (including earring) in the next 60 days.
* Use of any prescription or non-prescription medication that could inhibit bone marrow or liver function.
* Any previous treatment with any interferon product.
* Participation in any other investigational drug study within the 4 weeks prior to Day 1 or within 5 half-lives of the investigational treatment, whichever is longer.
* Treatment with the Flu Vaccine within 1 week prior to Day 1.

NOTE: Other protocol-defined inclusion/exclusion Criteria May Apply

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 69 (Actual)
Dates: Start 2008-03; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
The number of participants that experience Adverse Events (AEs) | Up to Day 71
The number of participants that experience flu-like symptoms | Up to Day 71
Participant assessment of injection site pain as measured by scores on a scale of 0 to 10, where 0 is no pain and 10 is extremely painful. | Up to Day 71
Clinician assessment of the injection site for erythema as assessed by a scale 0 to 3, where 0 represents no erythema and 3 represents severe erythema | Up to Day 71
Clinician assessment of the injection site for induration as assessed by a scale 0 to 3, where 0 represents no induration and 3 represents severe induration | Up to Day 71
Clinician assessment of tenderness to digital pressure at the injection site will be assessed on a scale of 0 to 3, where 0 represents no tenderness and 3 represents severe tenderness | Up to Day 71
Clinician assessment of temperature at the injection site will be assessed on a scale of 0 to 2, where 0 represents normal temperature and 2 represents hot. | Up to Day 71

SECONDARY OUTCOMES:
AUC168h, area under the concentration-time curve | Up to 168 hours post dose
Cmax, observed maximum serum concentration | Up to 336 hours post-dose
Tmax, time to reach maximum serum concentration | Up to 336 hours post-dose
Terminal t½, half-life of the terminal phase | Up to 336 hours post-dose
EAUC-336h, area under the concentration-time curve from time zero to 336 hours post-dose | Up to 336 hours post-dose
Emax, the peak concentration observed minus baseline concentration | Day 1 and Day 29
PD parameters of serum concentrations of neopterin | Day 1 and Day 29

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (1):
- Research Site, Phoenix, Arizona, United States

REFERENCES:
- [Result] Hu X, Miller L, Richman S, Hitchman S, Glick G, Liu S, Zhu Y, Crossman M, Nestorov I, Gronke RS, Baker DP, Rogge M, Subramanyam M, Davar G. A novel PEGylated interferon beta-1a for multiple sclerosis: safety, pharmacology, and biology. J Clin Pharmacol. 2012 Jun;52(6):798-808. doi: 10.1177/0091270011407068. Epub 2011 Jun 16. PMID 21680782